CLINICAL TRIAL: NCT06875609
Title: ctDNA Clearance and ctDNA Monitoring Study in Cutaneous Squamous Cell Carcinoma
Brief Title: ctDNA in Cutaneous Squamous Cell Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Haystack Oncology, Inc. (Unknown); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sophia Shalhout, PhD, Assistant Professor, Massachusetts Eye and Ear Infirmary
Other Study IDs: 2024P003225
Record Dates: First submitted 2025-02-10; First posted 2025-03-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Cutaneous Squamous Cell Carcinoma
Keywords: Circulating Tumor DNA; CSCC; Skin cancer; Biomarker; ctDNA; Minimal Residual Disease (MRD); Liquid Biopsy; Advanced Skin Cancer
MeSH Terms: conditions — Skin Neoplasms; Neoplasm, Residual | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma and CSCC tumor tissue- Tumor biopsy specimens will be used to develop personalized ctDNA assay. Blood will be serially collected for ctDNA analysis. DNA is extracted from these tissues for assay development and assessment/analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post-Operative Cohort: Cutaneous Squamous Cell Carcinoma cancer patients treated with surgery.
  Interventions: Diagnostic Test: Blood and Tissue Collection
- Neoadjuvant Cohort: Cutaneous Squamous Cell Carcinoma patients treated with Neoadjuvant immunotherapy.
  Interventions: Diagnostic Test: Blood and Tissue Collection
- Definitive Immunotherapy Cohort: Cutaneous Squamous Cell Carcinoma patients treated with definitive immunotherapy.
  Interventions: Diagnostic Test: Blood and Tissue Collection

INTERVENTIONS:
Diagnostic Test: Blood and Tissue Collection — Blood samples, and tissue samples will be collected from the participants, and used to determine whether circulating tumor DNA (ctDNA) testing can help monitor treatment in patients with CSCC, and to determine how ctDNA levels change in patients.
  Other Names: ctDNA test

SUMMARY:
The purpose of this study is to test the potential for a liquid biopsy assay to detect residual disease after surgery in patients with cutaneous squamous cell carcinoma as well as the potential for this assay to monitor response to immunotherapy treatment.

DETAILED DESCRIPTION:
The study aims to better understand whether circulating tumor DNA, or ctDNA, a type of personalized blood test informed by the tumor, can help monitor recurrence and treatment responses in patients with cutaneous squamous cell carcinoma (CSCC), especially during and after treatment. Blood samples will be collected during regular treatment visits or through mobile phlebotomy visits, and analyzed to study how ctDNA levels change over time. Participants will be in the study for 2 years.

Circulating tumor DNA consists of small fragments of DNA shed into the bloodstream by cancer cells. It may serve as a non-invasive biomarker for detecting and monitoring CSCC, offering insights into tumor treatment response and/or progression. ctDNA can provide a "liquid biopsy," allowing real-time tracking of tumor dynamics. Specifically, the study is researching how ctDNA levels change in patients undergoing surgery, immunotherapy, or other standard treatments. The goal is to see if ctDNA can serve as a biomarker to better understand treatment response and detect potential progression/ recurrence of the cancer.

This study does not involve any experimental drugs or devices. All drugs and treatments administered to participants, including surgery and immunotherapy, are part of standard of care. The ctDNA blood test is being used as a research tool and is not currently approved by the U.S. Food and Drug Administration (FDA) for monitoring CSCC. The study aims to evaluate its potential future use as a reliable biomarker.

ELIGIBILITY:
Post-Operative Cohort

Inclusion Criteria:

* Patients with surgically resectable primary CSCC with PNI (>0.1mm caliber nerve) or at least 2 high-risk features defined as size > 2cm, recurrent CSCC, LVI, immunosuppressed, poorly differentiated, and/or invasion >6mm/beyond subcutaneous fat;
* Patients with surgically resectable regional metastases not receiving neoadjuvant therapy

Exclusion Criteria:

* Patients with Cutaneous Squamous Cell Carcinoma not amenable to surgical resection
* Patients receiving or undergoing systemic therapies.

Neoadjuvant Cohort

Inclusion Criteria:

* Patients with resectable AJCC (8th ed) Stage II, III or IV(M0) CSCC treated with neoadjuvant immunotherapy as part of standard care.

Exclusion Criteria:

* Patients ineligible for neoadjuvant treatment.

Definitive Immunotherapy Cohort

Inclusion Criteria:

* Patients with unresectable locally advanced or metastatic CSCC, AJCC (8th ed) Stage II, III, or IV), receiving immunotherapy as part of standard of care.

Exclusion Criteria:

* Patients undergoing systemic therapies outside the standard of care or enrolled in conflicting clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ages 18 and older, who have been diagnosed with cutaneous squamous cell carcinoma (CSCC)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
2-year recurrence-free survival (RFS) in patients with detectable vs no detectable ctDNA after surgery | 24 Months
  To determine if there is an association between ctDNA clearance (defined as no detection of ctDNA) after surgical intervention and 2-year recurrence-free survival (RFS). The outcome will measure both ctDNA clearance (as a binary variable: detection or no detection) and RFS (measured in months). The association between these two outcomes will be analyzed as the primary outcome to determine if no detection of ctDNA is associated with longer RFS.
Neoadjuvant Cohort Primary Outcome: Response Monitoring | 24 Months
  To evaluate ctDNA as a biomarker of response to neoadjuvant immunotherapy.
Definitive Treatment Cohort Primary Outcome | 24 Months
  To evaluate whether ctDNA correlates with response to immunotherapy.

SECONDARY OUTCOMES:
Post-Operative Cohort Secondary Outcome: Residual Free Survival (RFS) Surveillance over 2 Year | 24 Months
  To evaluate RFS during the surveillance period, stratified by ctDNA test status over time to determine if ctDNA levels predict recurrence
Neoadjuvant Cohort Secondary Outcome: Correlation with Pathological Response | 24 Months
  To evaluate if ctDNA correlates with pathological response to neoadjuvant therapy. This will help determine if ctDNA may one day be used to help risk stratify which patients need surgery after neoadjuvant immunotherapy.

OTHER OUTCOMES:
Exploratory Outcome | 24 Months
  To evaluate the time to ctDNA clearance (defined as the time from surgical intervention to the point where ctDNA is no longer detected, if ever) in the postoperative period, defined as months since surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Z. Shalhout, PhD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No